CLINICAL TRIAL: NCT03627975
Title: Effect of Surgical Revascularization and Conservative Treatment on Hemorrhagic Moyamoya Disease
Brief Title: Effect of Surgical Revascularization on Hemorrhagic Moyamoya Disease
Acronym: ESRHMMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z171100001017144
Record Dates: First submitted 2018-07-29; First posted 2018-08-14 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Moyamoya Disease
Keywords: revascularization; hemorrhagic moyamoya disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative treatment (No Intervention): Conservative treatment. The conservative treatment of hemorrhagic moyamoya disease mainly includes the control of hypertension, the prevention and treatment of secondary epilepsy, the control of intracranial hypertension(including the application of mannitol and glycerol fructose, etc.), and the corresponding symptomatic and neurotrophic treatment. Non-specific treatment is mainly deal with intracranial hematoma, including intraventricular drainage, intracranial hematoma evacuation, and ventriculoperitoneal shunt.
- Indirect vascular reconstruction surgery (Experimental): Indirect vascular reconstruction surgery. In addition to the pharmacotherapy used in conservative treatment, encephalo-duro-arterio-synangiosis(EDAS) is performed. The surgery is performed according to the procedures described by Matsushima.
  Interventions: Procedure: Conservative treatment
- direct vascular reconstruction surgery (Experimental): Direct vascular reconstruction surgery. In addition to the pharmacotherapy used in conservative treatment, the superficial temporal artery(STA) and middle cerebral artery(MCA) bypass surgery is performed. The operation is the modified EDAS which basically similar to EDAS, but the surgical incision is as low as possible. And if necessary, the STA may not be preserved. The bone flap should be large enough to select the right recipient blood vessel.
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Conservative treatment — 1. The conservative treatment of hemorrhagic moyamoya disease mainly includes the control of hypertension, prevention and treatment of secondary epilepsy, the control of intracranial hypertension, and the corresponding symptomatic and neurotrophic treatment.
  2. In addition to the pharmacotherapy used in conservative treatment, encephalo-duro-arterio-synangiosis(EDAS) will be performed according to the procedures described by Matsushima.
  3. In addition to the pharmacotherapy used in conservative treatment, the superficial temporal artery(STA) and middle cerebral artery(MCA) by pass surgery is performed. The operation is the modified EDAS which basically similar to EDAS, but the surgical incision is as low as possible. And the STA may not be preserved.
  Other Names: indirect revascularization; direct revascularization
  Arms: Indirect vascular reconstruction surgery; direct vascular reconstruction surgery

SUMMARY:
Moyamoya Disease(MMD), also known as spontaneous basilar artery occlusion, is characterized by the gradual thickening of arterial intima at the distal carotid artery and the proximal portion of anterior/middle cerebral artery, the gradual stenosis or occlusion of arterial lumen, and the compensatory expansion of basilar cerebral perforating arteries. Cerebral infarction and cerebral hemorrhage are common clinical symptoms of MMD with high morbidity of disability. For ischemic moyamoya disease, intracranial/extracranial revascularization is the preferred treatment. However, for patients with hemorrhagic moyamoya disease, there is controversy about whether to have surgical treatment, the timing and the method of surgical treatment, and the effect of surgical treatment to prevent rebleeding due to the lack of large sample, multi-center, prospective randomized studies. At present, the studies on the effect of revascularization and conservative treatment on hemorrhagic moyamoya disease are retrospective case analyses without randomized control. The sample size of these studies are small, and the conclusions obtained are inconsistent. Due to the differences in the epidemiology and episode type of moyamoya disease in different countries, there is no prospective, randomized controlled study of blood type moyamoya disease in China to confirm the efficacy of revascularization and lack of uniform norms and standards.

DETAILED DESCRIPTION:
Objective: The aim of this study is to perform a prospective, randomized study on hemorrhagic moyamoya disease to confirm the effect of revascularization in China, and to establish specifications and standards to guide the treatment options for hemorrhagic moyamoya disease as well.

Design: This study is a single-center study and plan to include 108 patients. According to a random number table, hemorrhagic moyamoya patients will be assigned to three groups: conservative treatment group, direct revascularization group and indirect revascularization group. A prospective, randomized study will be carried out to evaluate the effect of revascularization and conservative treatment on the reduction of rebleeding risk and improvement of ischemia in adult patients with hemorrhagic moyamoya disease.

Observation Measures: 1.Rebleeding; 2.Cerebral infarction resulting in severe disability (mRS score≥3); 3.Severe disability or death caused by other reasons; 4. Patients in conservative treatment group need revascularization due to progressive ischemic stroke or progressive Transient ischemic attack(TIA).

ELIGIBILITY:
Inclusion Criteria:

* DSA/MRA shows stenosis or occlusion in the distal internal carotid artery or the proximal portion of anterior/middle cerebral artery
* Abnormal vascular network appeared in the brain
* Lesions showed bilateral changes
* Age≥18 years
* With the onset of cerebral hemorrhage
* No cerebral infarction or cerebral hemorrhage occurred within the last month
* At least one month after the acute phase of cerebral hemorrhage or related diseases was treated

Exclusion Criteria:

* Patients with moyamoya syndrome secondary to systemic diseases such as arteriosclerosis, sickle cell anemia, radiation therapy, etc..
* Patients with severe mental disorders such as psychosis, liver and kidney dysfunction, poor blood pressure or blood glucose control, severe depression and substance abuse, low IQ, and acute phase of severe stroke with definite limb dysfunction should also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | Through study completion, an average of 1 year
  All enrolled patients were followed up regularly by telephone, outpatient and inpatient visits. The observed end-point events of rebleeding

SECONDARY OUTCOMES:
Severe Disability | Through study completion, an average of 1 year
  Cerebral infarction resulting in severe disability (mRS score≥3)
Severe Disability or Death | Through study completion, an average of 1 year
  Severe disability or death caused by other reasons
Vascular Reconstruction due to Progressive Ischemic Stroke or Progressive TIA | Through study completion, an average of 1 year
  Patients in conservative treatment group needs vascular reconstruction due to progressive ischemic stroke or progressive TIA.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Lian, Chief, Study Chair — The 307th Hospital of Military Chinese People's Liberation Army
Locations (1):
- The 307th Hospital of Military Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No